CLINICAL TRIAL: NCT05336565
Title: Incidence of Prescribing Potentially Inappropriate Medications to Older Cardiovascular Patients During COVID-19 Pandemics According to Medical Information System BARS
Brief Title: PIM Incidence in Older Cardiovascular Patients During COVID-19 Pandemics
Acronym: PIM-BARS
Status: Recruiting | Type: Observational
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Responsible Party: Principal Investigator, Nina D. Anfinogenova, Leading Research Scientist, Tomsk National Research Medical Center of the Russian Academy of Sciences
Other Study IDs: PIM-BARS
Record Dates: First submitted 2022-04-19; First posted 2022-04-20 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Potentially Inappropriate Medications
Keywords: Potentially inappropriate medication; Drug-drug-interaction; Polypharmacy; Cardiovascular; Electronic medical record; Medical information system; Prevention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Electronic medical record analysis — Medical information system (MIS) "BARS" will be used for inclusion and retrieval of relevant data of cardiovascular patients enrolled in the reimbursement programs in the Tomsk Region. Incidence rates and patterns of PIM prescription, polypharmacy, and PDDIs in the time of COVID-19 pandemic will be studied.

SUMMARY:
The aim of the study is to assess the incidence of potentially inappropriate medication (PIM) administration, polypharmacy, and potential drug-drug-interactions (PDDIs) in cardiovascular patients enrolled in the reimbursement program in the time of coronavirus disease (COVID-19) pandemic. Medical information system (MIS) "BARS" will be used for inclusion and retrieval of relevant data of cardiovascular patients enrolled in the reimbursement programs in the Tomsk Region. The incidence rates of PIM prescriptions will be assessed in patients aged 75 years and older. Potentially inappropriate medications will be defined according to 2015 Beers criteria. Polypharmacy will be defined as being administered five or more medications at the same time. PDDIs will be checked with Medscape Drug Interaction Checker and rated as 'Contraindicated', 'Serious', and 'Requiring Monitoring'. Combined analysis of retrospective and prospective occurrences of study parameters will be performed. PIM-BARS will evaluate the incidence rates and patterns of PIM prescriptions, polypharmacy, and PDDIs in elderly cardiovascular patients enrolled in the reimbursement program in the time of COVID-19 pandemic.

DETAILED DESCRIPTION:
Objective: It is essential to improve patient safety by determining an individual's exposure to potentially inappropriate drugs.

This study will be performed to find out the incidence of potentially inappropriate medication (PIM) administration, polypharmacy, and potential drug-drug-interactions (PDDIs) in cardiovascular patients enrolled in the reimbursement program in the time of COVID-19 pandemic.

Method: Medical information system (MIS) "BARS" will be used for inclusion and retrieval of relevant data of cardiovascular patients enrolled in the reimbursement programs in the Tomsk Region. Incidence of PIM administration, polypharmacy, and PDDIs in the time of COVID-19 pandemic will be studied. Brief characteristics of MIS "BARS" implemented in the Diagnostic and Consultation Center of Cardiology Research Institute, Tomsk National Research Medical Center, Russian Academy of Sciences (NRMC) are as follows: MIS "BARS" is a universal solution for automatization of activities of medical institutions of various specializations and scale ranging from small highly specialized clinics to multi-specialty hospitals and medical centers. The system is the united information space for administrative, treatment-and-diagnostic, and financial-and-economic processes of medical institution. MIS "BARS" is a cloud-based solution, and the deployment of the system in cloud allows getting the remote access to working places from any location. The system is built based on module principle. The system implements automatic control over provision of medical services allowing for feedback with practical healthcare workers. The system is integrated with other information systems and medical equipment. The advantage of the system consists in a capability to assess economic element of study parameters. Technical characteristics of MIS "BARS": The system has a centralized data base with provision of protected remote access for users. The system is organized based on principle of three-tiered architecture: Web browser, Web-server, and database server. ORACLE is used as a database server, which provides the highest data security, scalability, fall-over protection, and the greatest capabilities for integration. Built-in mechanisms of functional system expansion allow to perform advanced customization.

Expected Results: Patient demographics, clinical data, instrumental examination data, and medication prescriptions will be collected using electronic medical records stored in medical information system (MIS) "BARS". The incidence rates of PIM prescriptions will be assessed. Potentially inappropriate medications will be defined according to 2015 Beers criteria. Polypharmacy will be defined as being administered five or more medications at the same time. PDDIs will be checked with Medscape Drug Interaction Checker and rated as 'Contraindicated', 'Serious', and 'Requiring Monitoring'. Combined analysis of retrospective and prospective occurrences of study parameters will be performed.

Conclusion: PIM-BARS will evaluate the incidence rates and patterns of PIM prescriptions, polypharmacy, and PDDIs in elderly cardiovascular patients enrolled in the reimbursement program in the time of COVID-19 pandemic. This effort will contribute to prevention of medication errors by inappropriate prescribing.

ELIGIBILITY:
Inclusion Criteria:

* established diagnosis of cardiovascular disease
* age of 18 years and older
* enrollment in the reimbursement program in Tomsk Region

Exclusion Criteria:

* age of 17 years and younger

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiovascular patients enrolled in the reimbursement program in Tomsk Region who have electronic medical records stored in medical information system BARS.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of potentially inappropriate medication prescription | Five years
  Incidence rate of potentially inappropriate medication prescriptions (PIM) will be assessed as annual percentage (%) of patient visits to medical doctors resulting in PIM prescription registered in medical information system BARS.

SECONDARY OUTCOMES:
Potential drug-drug interactions (PDDIs) | Five years
  Potential drug-drug interactions (PDDIs) will be checked with Medscape Drug Interaction Checker, rated as 'Contraindicated', 'Serious', and 'Requiring Monitoring', and assessed as percentage (%) of patients exposed to them based on data of medical information system BARS.
Polypharmacy rate | Five years
  Polypharmacy is defined as being prescribed five or more medications at the same time and assessed as percentage (%) of patients exposed to it based on data of medical information system BARS.

CONTACTS AND LOCATIONS:
Overall Officials: Nina D Anfinogenova, MD, PhD, Principal Investigator — Cardiology Research Institute, Tomsk National Research Medical Center, Russian Academy of Sciences; Alexey N Repin, MD, PhD, Study Director — Cardiology Research Institute, Tomsk National Research Medical Center, Russian Academy of Sciences
Locations (1):
- Tomsk NRMC, Tomsk, Russia

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data (text, tables, figures, and appendices), underlying the results of the trial, will be shared with researchers to achieve the aims in the approved proposal.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Proposals may be submitted up to 36 months following publication of the results of the trial. After 36 months, the data will be available in the Center's data ware house but without investigator support other than deposited metadata.
Access Criteria: Information regarding submitting proposals and accessing data may be requested from the principal investigator by e-mail.